CLINICAL TRIAL: NCT03975582
Title: Somnotouch-NIBP Compared to Standard Ambulatory 24 Hours Blood Pressure Measurement - a Prospective Registry
Brief Title: Somnotouch-NIBP Compared to Standard Ambulatory 24-hours Blood Pressure Measurement
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: VAST-Registry
Record Dates: First submitted 2019-04-24; First posted 2019-06-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison of 24 hours blood pressure measurement with puls-transit time versus cuffs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to give informed consent

Exclusion Criteria:

* Age < 18 years
* Medical reasons that forbid blood pressure measurements on upper extremities
* Not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the medical outpatient clinic of the University Hospital of Basel with an indication for an ambulatory 24h blood pressure measurement.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in mean 24 hours systolic blood pressure | 24 hours
  Difference in mean 24 hours systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Burkard, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derendinger FC, Vischer AS, Krisai P, Socrates T, Schumacher C, Mayr M, Burkard T. Ability of a 24-h ambulatory cuffless blood pressure monitoring device to track blood pressure changes in clinical practice. J Hypertens. 2024 Apr 1;42(4):662-671. doi: 10.1097/HJH.0000000000003667. Epub 2024 Jan 23. PMID 38288945